CLINICAL TRIAL: NCT05512117
Title: Análisis de la utilización de Los catéteres Intravenosos periféricos de Linea Media Frente a Los catéteres Intravenosos periféricos Convencionales en el Servicio de Medicina Interna
Brief Title: Midline Catheters Versus Peripheral Catheters in Internal Medicine Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Elena Chover Sierra, Principal Investigator, Hospital General Universitario de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HGUValencia_midline
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Vascular Access Complication; Vascular Access Device Complications
Keywords: phlebitis
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: Intravenous access catheter in control group is conventional intravenous catheter (Braun Introcan Safety) Intravenous access catheter in intervention group is a midline catheter 12 cm length (Leader Cath 20 G. Vygon)
Who Masked: Outcomes Assessor
Masking Description: Neither care providers nor patients could be masked because the intravenous device is different and it's easy to identify the one we are using.
  Outcomes assessor only works with anonymized data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midline Catheter (Experimental): Midline catheter insertion
  Interventions: Device: Midline insertion
- Peripheral intravenous cannulation (PIVC) (No Intervention): Peripheral intravenous cannulation (PIVC)

INTERVENTIONS:
Device: Midline insertion — Midline catheter insertion
  Arms: Midline Catheter

SUMMARY:
The study aims to evaluate the rate of complications and the duration of cannulation of a midline intravenous catheter compared to a short peripheral catheter in patients hospitalized in an Internal Medicine service of a Spanish hospital.

DETAILED DESCRIPTION:
A randomized, longitudinal experimental study is designed, which will allow comparisons to be made between the results obtained in the experimental group and the control group.

The study will be carried out in the Internal Medicine and medium and long stay unit of the CHGUV, during the period of time necessary to complete the required sample size, which has finally been established at six months.

When the patient is admitted to our unit, a number is assigned from the admission service, based on their admission order; this number will serve for subsequent random assignment to one another group. In this case, the use of a website to generate said numbers is proposed.

Using established procedures for the generation of random numbers, the numbers that correspond to the subjects that are going to be part of each of the groups will be identified.

The list of random numbers that will make up the experimental group has been prepared previously by the Internal Medicine Unit secretary and will be known by the person who will carry out the placement of the midline catheter (two nurses from the unit trained in the placement and handling of this type of device, who will also be those in charge of training the rest of the staff).

The list will be reviewed daily in the morning shift, and those patients who have not given their informed consent will be eliminated, those in whom, due to their pathology, a brief admission is expected or patients who are in a terminal or palliative care situation, in those who consider the step of treatment to the subcutaneous route as the best option.

The informed consent to participate in the study will be given to the patient and/or relatives at the time of admission, also informing them that the next morning those responsible for the study will explain the object of the study in more depth and answer their questions.

Before the third day after admission, in the morning shift, the peripheral catheters will be reviewed and replaced by another peripheral catheter or by a midline catheter depending on the group to which the patient has been assigned. In case of being a patient assigned to the experimental group, the midline catheter will be placed by personnel trained for it.

The procedures for inserting and maintaining the catheters are already established in the unit and will be those that will be followed during the study, depending on the type of catheter; The care in the insertion and maintenance of midline catheters does not differ from the care of peripherally inserted central catheters, since they require a sterile technique; therefore, although the insertion of the midline catheters will be done by the selected investigators, maintenance will be performed by the unit's staff, following, as we have indicated, the procedures already established.

When the patient requires a change of venous access for whatever reason, it will be replaced by the same type of catheter (midline or conventional catheter) and the necessary information will be added to the information record sheet.

ELIGIBILITY:
Inclusion Criteria:

* The patients included were those who were hospitalized in the Internal Medicine Service of the Consorcio Hospital General Universitario de Valencia who needed intravenous therapy and who had signed the Informed Consent for placement of a midline at the time of the change of the PIVC placed in the emergency unit.

Exclusion Criteria:

* Those with a forecast hospitalization of less than one week, those who were receiving palliative or symptomatic treatment, those who were carriers of a CVC or those who had presented difficulty in venous access with midline after two consecutive attempts were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Length of canalization | Four weeks
  Days of catheter stay
Number of punctures | Four weeks
  Number of times a catheter is inserted
Phlebitis | Four weeks
  Presence of catheter related phlebitis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Millington SJ, Hendin A, Shiloh AL, Koenig S. Better With Ultrasound: Peripheral Intravenous Catheter Insertion. Chest. 2020 Feb;157(2):369-375. doi: 10.1016/j.chest.2019.04.139. Epub 2019 Oct 22. PMID 31654617
- [Background] Prasanna N, Yamane D, Haridasa N, Davison D, Sparks A, Hawkins K. Safety and efficacy of vasopressor administration through midline catheters. J Crit Care. 2021 Feb;61:1-4. doi: 10.1016/j.jcrc.2020.09.024. Epub 2020 Oct 2. PMID 33049486
- [Background] Nickel B. Does the Midline Peripheral Intravenous Catheter Have a Place in Critical Care? Crit Care Nurse. 2021 Dec 1;41(6):e1-e21. doi: 10.4037/ccn2021818. PMID 34851379
- [Background] Moureau N, Chopra V. Indications for peripheral, midline and central catheters: summary of the MAGIC recommendations. Br J Nurs. 2016 Apr 28-May 11;25(8):S15-24. doi: 10.12968/bjon.2016.25.8.S15. PMID 27126759
- [Background] Skaggs MKD, Daniels JF, Hodge AJ, DeCamp VL. Using the Evidence-Based Practice Service Nursing Bundle to Increase Patient Satisfaction. J Emerg Nurs. 2018 Jan;44(1):37-45. doi: 10.1016/j.jen.2017.10.011. Epub 2017 Nov 20. PMID 29167032
- [Background] Mohn-Brown E. Implementing Quality and Safety Education for Nurses in Postclinical Conferences: Transforming the Design of Clinical Nursing Education. Nurse Educ. 2017 Sep/Oct;42(5S Suppl 1):S18-S21. doi: 10.1097/NNE.0000000000000410. PMID 28832457
- [Background] Johansen H, Helgesen AK. Palliative care in the community - the role of the resource nurse, a qualitative study. BMC Palliat Care. 2021 Oct 14;20(1):157. doi: 10.1186/s12904-021-00860-w. PMID 34645424
- [Background] Selby LM, Rupp ME, Cawcutt KA. Prevention of Central-Line Associated Bloodstream Infections: 2021 Update. Infect Dis Clin North Am. 2021 Dec;35(4):841-856. doi: 10.1016/j.idc.2021.07.004. PMID 34752222
- [Background] Panepinto R, Harris J, Wellette J. A Review of Best Practices Related to Intravenous Line Management for Nurses. Nurs Clin North Am. 2021 Sep;56(3):389-399. doi: 10.1016/j.cnur.2021.05.001. PMID 34366159
- [Background] Timsit JF, Baleine J, Bernard L, Calvino-Gunther S, Darmon M, Dellamonica J, Desruennes E, Leone M, Lepape A, Leroy O, Lucet JC, Merchaoui Z, Mimoz O, Misset B, Parienti JJ, Quenot JP, Roch A, Schmidt M, Slama M, Souweine B, Zahar JR, Zingg W, Bodet-Contentin L, Maxime V. Expert consensus-based clinical practice guidelines management of intravascular catheters in the intensive care unit. Ann Intensive Care. 2020 Sep 7;10(1):118. doi: 10.1186/s13613-020-00713-4. PMID 32894389
- [Background] Farina J, Cornistein W, Balasini C, Chuluyan J, Blanco M. [Central venous catheter related infections. Inter-Societies update and recommendations]. Medicina (B Aires). 2019;79(1):53-60. Spanish. PMID 30694189
- [Background] Scoppettuolo G, Pittiruti M, Pitoni S, Dolcetti L, Emoli A, Mitidieri A, Migliorini I, Annetta MG. Ultrasound-guided "short" midline catheters for difficult venous access in the emergency department: a retrospective analysis. Int J Emerg Med. 2016 Dec;9(1):3. doi: 10.1186/s12245-016-0100-0. Epub 2016 Feb 4. PMID 26847572
- [Derived] Villalba-Nicolau M, Chover-Sierra E, Saus-Ortega C, Ballestar-Tarin ML, Chover-Sierra P, Martinez-Sabater A. Usefulness of Midline Catheters versus Peripheral Venous Catheters in an Inpatient Unit: A Pilot Randomized Clinical Trial. Nurs Rep. 2022 Oct 31;12(4):814-823. doi: 10.3390/nursrep12040079. PMID 36412798
- Available data/document: Study Protocol — https://www.uv.es/uvweb/servei-investigacio/ca/grups-investigacio/grup-1285949714098.html?p2=GIUV2019-456 — All study information can be requested via email.